CLINICAL TRIAL: NCT00293657
Title: A Randomized, Double-Blind, Single-Dose Study, Placebo-Controlled Evaluation of the Safety and Efficacy of Intravenous Lornoxicam in the Acute Treatment of the Headache of Migraine.
Brief Title: Study of Lornoxicam or Placebo for Acute Treatment of the Headache of Migraine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POZEN (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNP-201
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Headache (Migraine)
MeSH Terms: conditions — Migraine Disorders | interventions — lornoxicam

INTERVENTIONS:
Drug: Lornoxicam 8 mg
Drug: Lornoxicam 16 mg
Drug: Placebo

SUMMARY:
To determine whether a single dose of intravenous lornoxicam is superior to intravenous placebo for the acute treatment of moderate or severe headache associated with a single migraine attack in patients with a history of migraine. Two-thirds of patients in this study will receive a single dose of intravenous lornoxicam (8mg or 16 mg) and one-third of patients will receive a single dose of an intravenous placebo.

DETAILED DESCRIPTION:
The headache of migraine is the primary symptom of this disorder that is estimated to affect approximately 10% of the population of developed countries, with the majority of persons with migraine being females between the ages of 20 and 50 years. Patients with migraine desire rapid and complete relief from headache and decreased frequency of recurrence over the 24 hours after treatment. Current treatments for migraine often provide incomplete pain relief and additional acute treatments are needed. Lornoxicam is a member of the NSAID class of anti-inflammatory drugs and is shown to be effective in the acute management of postoperative pain and arthritis. The current study will evaluate the efficacy of single doses of lornoxicam, administered intravenously, in treatment of the headache of migraine to determine possible future uses of this drug in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a demonstrated history of migraine headaches according to the International Headache Society (IHS) criteria 1.1 or 1.2 (2004), had their first migraine prior to age 50, and have had an average migraine headache frequency of 2-6 migraines per month, of moderate or severe pain intensity, in each of the last 6 months prior to screening.
* Subjects are willing to come to the study site when he/she has onset of the headache of migraine to receive an intravenous dose of study medication and is willing to remain in the investigator's clinic for at least 2 hours after the intravenous dose for collection of study data (Subject is discharged to home after 2 hour post-dose evaluations are completed).

Exclusion Criteria:

* Subjects who are pregnant.
* Subjects has known allergic reactions or intolerance to NSAIDs; any subject in whom aspirin or other non-steroidal anti-inflammatory/analgesic drugs induce the symptoms of asthma, rhinitis and nasal polyps.
* Subject is receiving any medications known or suspected to have drug interactions with lornoxicam. These include: warfarin or other anticoagulants, digoxin, probenecid, methotrexate, lithium, aspirin, cimetidine, cyclosporine and/or furosemide.
* Subjects with a non-migraine (i.e., tension-type, sinus, etc.) headache frequency of >15 days/month in each of the 3 months (90 days) prior to screening.
* Subjects experiencing greater than an average of 6 migraine attacks per month and/or >15 migraine days per month in the 6 months prior to screening.
* Subjects with a history of documented gastrointestinal ulceration in the past six months or hospitalization for gastrointestinal bleeding in the past year.
* Subjects with history of impaired renal function and/or a history of kidney disease, interstitial nephritis, nephrotic syndrome, and/or peripheral edema.
* Subjects with history of heart disease or certain related conditions.
* Subjects with uncontrolled hypertension or hypertension that is difficult to control with medications.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Assessment of headache pain intensity over 24 hours after treatment, rated on a categorical scale of 0-3 and a visual analog scale (VAS).

SECONDARY OUTCOMES:
Assessments of symptoms of photophobia, phonophobia, nausea and vomiting, rated as present or absent; use of rescue medication in the 24 hours after dosing; response of allodynia symptoms present at time of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James Adelman, MD, Principal Investigator — Headache Wellness Center; Sheena Aurora, MD, Principal Investigator — Swedish Pain Center; Gary Berman, MD, Principal Investigator — Clinical Research Institute; Roger Cady, MD, Principal Investigator — Headache Care Center; Merle Diamond, MD, Principal Investigator — Diamond Headache Clinic; Mildred Farmer, MD, Principal Investigator — Meridien Research; Gregory Flippo, MD, Principal Investigator — Alabama Clinical Therapeutics; Kevin Kahn, MD, Principal Investigator — University Headache Center; David Kudrow, MD, Principal Investigator — California Medical Clinic for Headache; Craig LaForce, MD, Principal Investigator — North Carolina Clinical Research; Ninan Mathew, MD, Principal Investigator — The Houston Headache Clinic; S. David Miller, MD, Principal Investigator — NE Medical Research Associates, Inc.; C. Phillip O'Carroll, MD, Principal Investigator — C. Phillip O'Carroll, MD, Inc.; Gilbert Podolsky, MD, Principal Investigator — Jean Brown Research; Kevin Roberts, MD, Principal Investigator — Little Rock Family Practice Clinic; John Rothrock, MD, Principal Investigator — University of South Alabama Neurology; Todd Rozen, MD, Principal Investigator — Michigan Head Pain and Neurological Institute; Stephan Sharp, MD, Principal Investigator — Clinical Research Associates, Inc.; Fred Sheftell, MD, Principal Investigator — New England Center for Headache; Stephen Silberstein, MD, Principal Investigator — Jefferson Headache Center; Timothy Smith, MD, Principal Investigator — Mercy Health Research / Ryan Headache Center; Stuart Stark, MD, Principal Investigator — The Innovative Clinical Research Center; Paul Winner, DO, Principal Investigator — Premiere Research Institute
Locations (23):
- United States (23):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - University of South Alabama Neurology, Mobile, Alabama
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - C. Phillip O'Carroll, MD, Inc., Newport Beach, California
  - California Medical Clinic for Headache, Santa Monica, California
  - New England Center for Headache, Stamford, Connecticut
  - Meridien Research, St. Petersburg, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - NE Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - Headache Care Center, Springfield, Missouri
  - Mercy Health Reserach / Ryan Headache Center, St Louis, Missouri
  - University Headache Center, Chapel Hill, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Jefferson Headache Center, Philadelphia, Pennsylvania
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Houston Headache Clinic, Houston, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - The Innovative Clinical Research Center, Alexandria, Virginia
  - Swedish Pain Center, Seattle, Washington